CLINICAL TRIAL: NCT04659096
Title: Phase 1 Trial of ION537 in Patients With Molecularly Selected Advanced Solid Tumors
Brief Title: A Study of ION537 in Patients With Molecularly Selected Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ionis Pharmaceuticals, Inc. (Industry)
Collaborators: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ION537-CS1
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Advanced Solid Tumors
Keywords: Solid tumors; Advanced solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- ION537 (Experimental): Multiple ascending doses of ION537 will be administered by intravenous (IV) injection on Days 1, 4, 8, 11, 15, and 22 in Cycle 1 and weekly dosing in each subsequent cycle until disease progression.
  Interventions: Drug: ION537

INTERVENTIONS:
Drug: ION537 — ION537 will be administered by IV injection.

SUMMARY:
The purpose of this study is to evaluate the safety and establish the maximum tolerated dose (MTD) and recommended Phase 2 dose (RP2D) of ION537 when administered by intravenous infusion in patients with advanced solid tumors.

DETAILED DESCRIPTION:
This is a single center, open label, non-randomized, Phase 1, two-part study of ION537 in up to 102 participants. Part 1 of the study consists of sequential cohort, dose escalation in patients with advanced solid tumors. Part 2 is dose expansion in patients with molecularly selected advanced solid tumors. In total, the study includes up to 102 participants. The study will consist of a 30-day screening period, a treatment period consisting of sequential consecutive treatment cycles (each cycle will be of 28 days) and a post-treatment follow-up period of at least 28 days following the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 18 years old
2. Participants must have histological diagnosis of local advanced (primary or recurrent) or metastatic solid tumors that are not amenable for treatment with curative intent
3. Participants must be in need of systemic treatment for their cancer and either are refractory to or have failed treatment with, are intolerant to or have refused, or are not otherwise a candidate, in the opinion of the Investigator, for any of the currently available established therapies
4. Participants must have available a fresh or recent tumor tissue sample from a diagnostic biopsy/surgery or a metastatic tumor biopsy;
5. Participants must have measurable disease by response evaluation criteria in solid tumors (RECIST) v1.1; or participants may have bone metastatic disease evaluable by Prostate Cancer Working Group 2 (PCWG2) for participants with metastatic castration-resistant prostate cancer (mCRPC), or according to the tumor evaluation criteria best suited and accepted for the tumor type being evaluated
6. Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
7. Participants must be willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other specified study procedures

Exclusion Criteria:

1. Known history or positive test for human immunodeficiency virus (HIV), hepatitis C virus (HCV) or chronic hepatitis B virus (HBV) infection.
2. Active infection requiring intravenous (IV) antibiotics
3. History of cerebrovascular accident (CVA), myocardial infarction or unstable angina within the previous 6 months before starting therapy.
4. Participants with uncontrolled Type I or II diabetes mellitus (DM); uncontrolled DM
5. Participants with prior anti-cancer therapy within 2 weeks prior to study enrollment or prior radiation therapy within 2 weeks prior to study enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-01-05 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE) and Treatment-emergent Serious Adverse Event (TESAE), Graded by Severity | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Number of Participants With Dose-limiting Toxicities (DLTs) | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Percentage of Participants With Complete Response (CR) | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Percentage of Participants With Partial Response (PR) | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Percentage of Participants With Stable Disease (SD) | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Area Under the Plasma Concentration-Time Curve from Hour Zero to Hour 24 AUC[0-24] for ION537 | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Maximum Observed Plasma Concentration (Cmax) for ION537 | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Inhibition of Yes-associated Protein (YAP1) Expression | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)

SECONDARY OUTCOMES:
Percentage of Participants With CR | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Percentage of Participants With PR | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Percentage of Participants With SD | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Clinical Benefit Rate (CBR) | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Objective Response Rate (ORR) | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Duration of Response (DoR) | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Progression-free Survival (PFS) | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Overall Survival (OS) | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Area Under the Plasma Concentration-Time Curve from Hour Zero to Hour 24 AUC[0-24] for ION537 | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Maximum Observed Plasma Concentration (Cmax) for ION537 | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Time to Reach the Maximum Plasma Concentration (Tmax) for ION537 | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)
Elimination Half-Life (t1/2) of ION537 | Up to disease progression, death, start of new anticancer treatment, withdrawal of consent to study participation or end of the study, whichever occurs first (up to approximately 24 weeks for analysis)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No